CLINICAL TRIAL: NCT00569192
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Study Investigating the Safety and Efficacy Over 12 Weeks Treatment Period of MAP0010 in Asthmatic Infants and Children 12 Months to 8 Years of Age
Brief Title: A Study of 2 Doses of MAP0010 and Placebo in Asthmatic Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAP0010-CL-P301
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: asthmatic children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.25mg MAP0010 (Experimental): 0.25mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 12 weeks
  Interventions: Drug: 0.25mg MAP0010
- Placebo (Placebo Comparator): Placebo delivered by nebulization twice daily for 12 weeks
  Interventions: Drug: Placebo
- 0.135mg MAP0010 (Experimental): 0.135mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 12 weeks
  Interventions: Drug: 0.135mg MAP0010

INTERVENTIONS:
Drug: 0.135mg MAP0010 — 0.135mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 12 weeks
  Arms: 0.135mg MAP0010
Drug: 0.25mg MAP0010 — 0.25mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 12 weeks
  Arms: 0.25mg MAP0010
Drug: Placebo — Placebo delivered by nebulization twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety and efficacy of two doses of MAP0010 versus placebo in asthmatic infants and children, 12 months to 8 years of age, over a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female asthmatic children with mild to moderate persistent asthma.
* 12 months to 8 years of age.
* For children age 4 to 8 years: Documented diagnosis of asthma at least 3 months prior to Visit 1, per NIH (EPR-3) criteria.
* For infants age 12 to <48 months old: 2 or more wheezing episodes in past 12 months which lasted > 1 day and affected sleep.
* AND with at least one major or two minor risk factors.

Exclusion Criteria:

* Any other significant childhood illness/abnormality or chronic lung disease
* Any history of upper or lower respiratory tract infection, within 2 weeks of screening.
* Any history of acute or severe asthma attack requiring ICU admission or ventilatory support.
* Use of any corticosteroid, including inhaled, parental, intranasal, or topical corticosteroid within 2 weeks of screening.
* Any use of oral corticosteroids within 30 days of screening or prolonged use (>10 consecutive days) of oral corticosteroids, within 12 weeks of screening.

Ages: 12 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — MAP Pharmaceuticals

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.135 mg MAP0010: 0.135mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 12 weeks
- 0.25 mg MAP0010: 0.125mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 12 weeks
Period: Overall Study
Arm/Group | Placebo | 0.135 mg MAP0010 | 0.25 mg MAP0010
Started | 111 | 125 | 124
Completed | 88 | 105 | 99
Not Completed | 23 | 20 | 25

BASELINE CHARACTERISTICS:
Groups:
- 0.25 mg MAP0010: 0.25mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.135 mg MAP0010 | 0.25 mg MAP0010 | Total
Number analyzed (Participants) | 111 | 125 | 124 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.5 (2.17) | 4.4 (2.33) | 4.2 (2.27) | 4.4 (2.26)
Age, Continuous [Median (Full Range); unit: years] | 4.0 [1 to 8] | 4.0 [1 to 8] | 4.0 [1 to 8] | 4.0 [1 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 49 | 144
  Male | 66 | 75 | 75 | 216

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daytime Composite Symptom Score
Description: The individual symptoms at each time point to be monitored are: cough, wheeze, and shortness of breath.
  The individual symptoms were scored using a four point scale:
  0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms
  Daily composite symptom score is based on the average of the individual symptom scores for a day. Daytime composite symptom score is defined as average of the last 5 days' daily composite symptom scores within the last 7 days immediately preceding the end day of that week. The range for the daytime composite symptom score is 0 (no symptoms) to 3 (severe symptoms). A negative change indicates an improvement of symptoms and a positive change indicates a worsening of symptoms.
Time Frame: baseline, week 12
Population: Intent-to-treat includes all randomized patients who have received at least one dose of study drug and have baseline and at least one post treatment efficacy assessment available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 0.135 mg MAP0010 | 0.25 mg MAP0010
Number analyzed (Participants) | 110 | 122 | 117
units on a scale
  Baseline | 2.73 (1.406) | 2.96 (1.329) | 2.87 (1.383)
  Change from Baseline at week 12 | -1.38 (1.722) | -1.77 (1.618) | -1.56 (1.591)

2. Secondary Outcome: Change From Baseline in FEV1% Predicted
Description: The forced expiratory volume in 1 second (FEV1) is the amount forced of air exhaled in 1 second. The percent predicted is calculated for age, gender, and height. Subjects had to perform at least 3 acceptable maneuvers into a spirometer and the largest volume from the 3 maneuvers was selected. An increase indicates an improvement (a greater volume of air expired).
Time Frame: baseline, week 12
Population: The modified-intent-to-treat population includes all randomized patients who were deemed capable of spirometry measurements at baseline and at least at one of the post treatment visits.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Placebo | 0.135 mg MAP0010 | 0.25 mg MAP0010
Number analyzed (Participants) | 38 | 37 | 40
percentage of predicted FEV1
  Baseline | 96.96 (18.646) | 91.20 (17.713) | 93.00 (17.305)
  Change from Baseline at Week 12 | 1.51 (13.068) | 4.14 (12.845) | 0.36 (16.657)

3. Primary Outcome: Change From Baseline in Nighttime Composite Symptom Score
Description: The individual symptoms at each time point to be monitored are: cough, wheeze, and shortness of breath.
  The individual symptoms were scored using a four point scale:
  0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms
  Nightly composite symptom score is based on the average of the individual symptom scores for the night. Nightime composite symptom score is defined as average of the last 5 days' nightly composite symptom scores within the last 7 nights immediately preceding the end day of that week. The range for the nighttime composite symptom score is 0 (no symptoms) to 3 (severe symptoms). A negative change indicates an improvement of symptoms and a positive change indicates a worsening of symptoms.
Time Frame: baseline, week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 0.135 mg MAP0010 | 0.25 mg MAP0010
Number analyzed (Participants) | 110 | 122 | 117
units on a scale
  Baseline | 2.71 (1.393) | 2.97 (1.466) | 2.82 (1.349)
  Change from Baseline at week 12 | -1.47 (1.572) | -1.82 (1.907) | -1.59 (1.516)

4. Secondary Outcome: Change From Baseline in PEF
Description: The peak expiratory flow (PEF) is the highest air flow achieved from a maximum forced expiratory maneuver measured in liters of air per minute (L/min). Subjects had to perform at least 3 acceptable maneuvers into a PEF meter. An increase indicates an improvement (a greater volume of air expired).
Time Frame: baseline, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Placebo | 0.135 mg MAP0010 | 0.25 mg MAP0010
Number analyzed (Participants) | 38 | 37 | 40
L/min
  Baseline | 170.94 (49.343) | 163.39 (52.881) | 165.34 (49.133)
  Change from Baseline at Week 12 | 0.71 (44.544) | 20.10 (45.444) | 15.02 (45.306)

5. Secondary Outcome: Change From Baseline in Daytime Individual Symptom Scores
Description: The individual symptoms at each time point to be monitored are: cough, wheeze, and shortness of breath.
  The individual symptoms were scored using a four point scale:
  0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms
  Individual Daytime symptom score is defined as an average of the last 5 days' individual symptom scores within the last 7 days immediately preceding the end day of that week. A negative change indicates an improvement of symptoms and a positive change indicates a worsening of symptoms.
Time Frame: baseline, week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 0.135 mg MAP0010 | 0.25 mg MAP0010
Number analyzed (Participants) | 110 | 122 | 117
units on a scale
  Cough: Baseline | 1.16 (0.544) | 1.21 (0.490) | 1.18 (0.582)
  Cough: Change from Baseline at week 12 | -0.55 (0.734) | -0.68 (0.705) | -0.58 (0.664)
  Wheeze: Baseline | 0.84 (0.591) | 0.91 (0.546) | 0.88 (0.550)
  Wheeze: Change from Baseline at week 12 | -0.45 (0.615) | -0.58 (0.563) | -0.49 (0.589)
  Shortness of Breath: Baseline | 0.73 (0.557) | 0.84 (0.612) | 0.81 (0.602)
  Shortness of Breath: Change from Baseline at Wk 12 | -0.37 (0.635) | -0.51 (0.632) | -0.49 (0.626)

6. Secondary Outcome: Change From Baseline in Nighttime Individual Symptom Scores
Description: The individual symptoms at each time point to be monitored are: cough, wheeze, and shortness of breath.
  The individual symptoms were scored using a four point scale:
  0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms
  Individual nighttime symptom score is defined as an average of the last 5 nights' individual symptom scores within the last 7 nights immediately preceding the end day of that week. A negative change indicates an improvement of symptoms and a positive change indicates a worsening of symptoms.
Time Frame: baseline, week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 0.135 mg MAP0010 | 0.25 mg MAP0010
Number analyzed (Participants) | 110 | 122 | 117
units on a scale
  Cough: Baseline | 1.16 (0.528) | 1.20 (0.495) | 1.17 (0.565)
  Cough: Change from Baseline at week 12 | -0.59 (0.663) | -0.69 (0.720) | -0.61 (0.638)
  Wheeze: Baseline | 0.83 (0.563) | 0.94 (0.592) | 0.90 (0.548)
  Wheeze: Change from Baseline at week 12 | -0.48 (0.594) | -0.57 (0.704) | -0.51 (0.603)
  Shortness of Breath: Baseline | 0.72 (0.543) | 0.83 (0.622) | 0.75 (0.569)
  Shortness of Breath: Change from Baseline at Wk 12 | -0.39 (0.549) | -0.56 (0.690) | -0.47 (0.566)

ADVERSE EVENTS:
Description: All randomized patients who received at least one dose of study drug and who have at least one post dosing safety evaluation were included in the adverse event analysis.
Arm/Group | Placebo | 0.135 mg MAP0010 | 0.25 mg MAP0010
Serious Adverse Events (participants affected / at risk) | 1/110 | 2/123 | 0/123
Other Adverse Events (participants affected / at risk) | 33/110 | 31/123 | 42/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=110) | 0.135 mg MAP0010 (N=123) | 0.25 mg MAP0010 (N=123)
Pneumonia Necrotising (Infections and infestations) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=110) | 0.135 mg MAP0010 (N=123) | 0.25 mg MAP0010 (N=123)
Pyrexia (General disorders) | 9 | 5 | 8
Upper Respiratory Tract Infections (Infections and infestations) | 13 | 17 | 19
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 15
Nasopharyngitis (Infections and infestations) | 5 | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.